CLINICAL TRIAL: NCT03634618
Title: Effects of Mirror Therapy After Carpal Tunnel Syndrome Surgery: Randomized Controlled Study
Brief Title: Efficiency of Mirror Therapy After Carpal Tunnel Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Tugba Karaaslan, Research Assistant, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IstanbulTK1
Record Dates: First submitted 2018-07-24; First posted 2018-08-16 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Carpal Tunnel Syndrome; Physiotherapy; Rehabilitation
Keywords: carpal tunnel syndrome; mirror therapy; postoperative rehabilitation; physical therapy modalities; median nerve
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Mirror Movement Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirror Therapy (Experimental): Mirror Therapy program for 2 weeks and convantional physiotherapy for 4 weeks. Exercises Frequency: 5 days/week; 2 days with the physiotherapist, other days as home program; 2 weeks in total. Exercises Duration: 20 minutes. Exercises Repetation: 20 repetation for each exercise.
  Interventions: Other: Mirror Therapy; Other: Convantional Physiotherapy
- Convantional Physiotherapy (Experimental): Convantional physiotherapy for 6 weeks. Exercises Frequency: 3 times a day, 4 weeks in total. Exercises Duration: 15-20 minutes. Exercises Repetation: 10 repetation for each exercise.
  Interventions: Other: Convantional Physiotherapy

INTERVENTIONS:
Other: Mirror Therapy — Mirror therapy is the treatment method in which mental performance of movements is performed by observing the movements of the healthy extremities. In the case of mirror treatment, the mirror box is placed on a fixed floor. The mirror is positioned so that the patient's body can be fully centered and the mirror image can be seen. While the affected limb is placed on the rear side of the mirror, the firm extremity is opposite to the mirror. The patient focuses on the mirror image of the moving healthy hand and, through artificial visual feedback, perceives the affected limb as moving. The exercises are as follows: flexor tendon gliding exercises, median motor exercises, wrist and forearm ROM exercises and function-oriented exercises.
  Arms: Mirror Therapy
Other: Convantional Physiotherapy — The first two weeks involve only immobilisation with plaster. The next 4 weeks, patients do the exercises which follows: 15 minutes water bath, scar tissue massage, flexor tendon gliding exercises, median motor exercises, wrist flexion-extention, median nerve gliding exercise (in addition, one week after plaster removal), hand wrist stretching exercise (in addition, 2 weeks after plaster removal).

SUMMARY:
In the randomized controlled study with patients who appropriate the inclusion criteria are divided into two groups by simple drawing method. In the control group, the classical physiotherapy program is being applied when the post-operative immobilization period ended, MT is applied to the mirror group in addition to this treatment for 20 minutes and a total of 10 sessions in the immobilization period. Patients who are scheduled for operation due to CTS evaluated that pain (VAS), sense (monofilament test), function (BCTQ, 9-hole peg test) before surgery, 3 weeks and 6 weeks after surgery.

DETAILED DESCRIPTION:
PURPOSE: The aim of this study is to investigate the efficacy of mirror therapy (MT).

METHOD: In the randomized controlled study with patients who appropriate the inclusion criteria are divided into two groups by simple drawing method. In the control group, the classical physiotherapy program is being applied when the post-operative immobilization period ended, MT is applied to the mirror group in addition to this treatment for 20 minutes and a total of 10 sessions in the immobilization period. Patients who are scheduled for operation due to CTS evaluated that pain (VAS), sense (monofilament test), function (BCTQ, 9-hole peg test) before surgery, 3 weeks and 6 weeks after surgery. The SPSS 21.0 statistical program will be used in the data analysis of the study and the level of significance wiil be accepted as p<0,05.

ELIGIBILITY:
Inclusion Criteria:

* Carpal tunnel diagnosis and open surgery are planned,
* Having the ability to adapt to exercises,
* Voluntarily agree to participate in the work

Exclusion Criteria:

* With the forearm and hand trauma story
* In the last 6 months, local corticosteroid injections to the treatment area have been performed
* Infection in the treatment area
* Having a deformity in hand
* The presence of malignancy
* Being pregnant

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2017-04-27 (Actual); Study Completion 2017-06-08 (Actual)

PRIMARY OUTCOMES:
Boston Carpal Tunnel Syndrome Questionnaire (the change of severity and functional status) | before surgery, 3 weeks and 6 weeks after surgery (3 repetitive measurements)
  It is a self-administered questionnaire that assesses the severity and functional status of typical 24-hour symptoms of patients with Carpal Tunnel Syndrome (CTS) during the last two weeks. The Symptom Severity Scale (SSS) consists of 11 questions evaluating the severity, frequency, duration and types of symptoms. The answers that can be given to each question are scored between 1 and 5. The SSS score is calculated by dividing the total score by the number of questions answered. A high score means that the symptoms are more severe. The Functional Status Scale (FSS) consists of 8 questions that assess how much the CTS affects daily life. The degree of difficulty in doing activities is scored between 1 and 5. The FSS score is calculated by dividing the total score by the number of questions answered. Higher score means less functional capacity.
  In this study, the outcome measure is assessing the change of functional activity and symptoms from pre-operative at 3 and 6 weeks.

SECONDARY OUTCOMES:
9-Hole Peg Test | before surgery, 3 weeks and 6 weeks after surgery
  It is used to evaluate patients' hand and finger skills. The pegboard is placed in the middle of the body. It is desirable that 9 wooden pins be placed randomly in the 9-hole wooden block as fast as possible, and then the pins are removed from the wooden block and placed in the storage compartment one by one. These times are measured and recorded with a stopwatch. A total of 20 seconds or more is considered a "loss of skill".
Semmes Weinstein Monofilaman Test | before surgery, 3 weeks and 6 weeks after surgery
  The sense of the distal phalanges of the 1st, 2nd and 3rd fingers, the proximal phalanges of the 2nd and 3rd fingers on the palm of the hand and the tenar region will be assessed. When the patient's eyes close, the monofilament is done progressed from the thinnest monofilament to the thicker monofilament, respectively. The assessment starts with the monofilament is perpendicular to the surface and pressure is applied until the angle is 45 degrees, wait for 1.5 seconds at this position. When at least 2 out of 3 applications differenciate, this value records.
Visual Analog Scale | before surgery, 3 weeks and 6 weeks after surgery
  The severity of pain and paresthesia symptoms of the patients will be assessed using the 10 cm Visual Analogue Scale. Before the assessment, patients instruct that "0" for "no symptoms", "10" represents "the most severe pain that could be felt" and should mark the point that best describes the symptom. The patient's rest, activity and night pain in the last week will be questioned separately. To evaluate the paresthesia, the most severe paresthesia felt by the patient in the last 1 week will be questioned and it will be asked to mark the place that best expresses paresthesia on the scale. Marked points measure by a ruler and record in centimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Tugba Karaaslan, Principal Investigator — Research Assistant
Locations (1):
- Istanbul University, Istanbul, Bakirkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No